CLINICAL TRIAL: NCT02466750
Title: Phase 2 Open-Label Safety and Immunogenicity Study of the Western Equine Encephalitis (WEE) Vaccine, Inactivated, Dried, TSI-GSD 210, Lot 3-1-92, in Healthy Adult Subjects at Risk of Exposure to Western Equine Encephalitis Virus
Brief Title: Safety and Immunogenicity Study of the Western Equine Encephalitis (WEE) Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-13-06
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Western Equine Encephalitis
MeSH Terms: conditions — Encephalomyelitis, Western Equine | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary vaccine (Experimental): Subjects receive 3 doses off WEE vaccine on Day 0, Day 7 ± 2 days, and Day 28-35 days. A booster will be administered on Day 180 ± 14 days and a sample collected for PRNT80 28-35 days later.
  Interventions: Biological: Western Equine Encephalitis (WEE) Vaccine
- Booster series (Experimental): Subjects who previously received the WEE vaccine under another protocol and have a PRNT80 < 1:40. Boosters (and follow-up titers 28-35 days later) may continue while the subject has titers of < 1:40 for a maximum of 4 booster doses in a year. If the titer remains < 1:40 after 4 booster doses in 1 year, the subject will not be given WEE vaccine for 1 year. If the titer is < 1:40 after that interval, one booster dose will be given and the titer will be assayed. If the immune response to the last booster dose is < 1:40, the subject will be considered to have completed the study as a nonresponder.
  Interventions: Biological: Western Equine Encephalitis (WEE) Vaccine

INTERVENTIONS:
Biological: Western Equine Encephalitis (WEE) Vaccine — Western Equine Encephalitis (WEE) Vaccine, Inactivated, Dried, TSI-GSD 210, Lot 3-1-92

SUMMARY:
This study is being conducted to collect safety and immunogenicity data for the WEE vaccine, TSI-GSD 210. Enrollment in this protocol is offered for personnel who enter areas where this virus is used in research or is endemic (an area where this disease process is found to occur frequently).

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 to 65 years old at time of consent.
2. Have WEE plaque reduction neutralization 80% titers (PRNT80) < 1:10 for primary series.
3. Have WEE PRNT80 < 1:40 for booster series.
4. If female of childbearing potential, must agree to have a urine pregnancy test on the same day before each vaccine. (Exception: documented hysterectomy or ≥ 3 years of menopause.) The results must be negative. Females must agree to not become pregnant for 3 months after receipt of the last study treatment (vaccination).
5. Be considered at risk for exposure to WEE virus and who have submitted a Request for IND Vaccines for the WEE vaccine.
6. Sign and date the approved informed consent document and HIPAA Authorization.
7. Have in their charts

   1. medical history (including concomitant medications) within 60 days of planned first administration of vaccine
   2. physical examination and laboratory tests within 1 year
   3. previous chest radiograph and electrocardiogram
8. Be medically cleared for participation by an investigator. (Examinations and/or tests may be repeated at the discretion of the enrolling physician.)
9. Be willing to return for all follow-up visits.
10. Agree to report any adverse events (AEs) that may or may not be associated with administration of the vaccine for at least 28 days after administration and agree to report all serious adverse events (for example, resulting in hospitalization) for the duration of the subject's participation in the study.
11. Agree to defer blood, bone marrow, and organ donation for 1 year after receipt of the vaccine.

Exclusion Criteria:

1. Have completed previous WEE vaccine study as a nonresponder (PRNT80 < 1:40).
2. Have clinically significant abnormal laboratory results (including evidence of hepatitis C, hepatitis B carrier state) or elevated liver function tests (two times the normal range or at the discretion of the PI).
3. Have a personal history of an immunodeficiency or received treatment with an immunosuppressive medication, such as systemically administered glucocorticoids (eg, prednisone) within 1 month before planned administration of the vaccine or with other immunosuppressive therapies within 6 months of planned administration of the vaccine. Other immunosuppressive therapies include all cancer chemotherapeutic agents, drugs to prevent transplant rejection, interferons, monoclonal antibodies, protein kinase inhibitors, methotrexate, TNF (tumor necrosis factor) inhibitors, and any other drug determined to be immunosuppressive by the PI. Current administration of topical, inhalational, or intranasal glucocorticoids is not excluded.
4. Have a confirmed HIV infection (antibody positivity).
5. Have a positive pregnancy test or be a breastfeeding female.
6. Have any known allergies to components of the vaccine:

   formaldehyde eggs neomycin sulfate human serum albumin sodium bisulfite
7. Have administration of another vaccine or investigational product within 28 days of WEE vaccination.
8. Have any unresolved AE resulting from a previous immunization.
9. A medical condition that, in the judgment of the PI, would impact subject safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-12-15 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | Up to 5 years
Percentage of subjects who develop titers of ≥ 1:40 as determined by PRNT80 | Up to 5 years
  Immunogenicity data will be collected for all subjects and will be evaluated for all per-protocol subjects. The primary immunogenicity endpoint measurements will be the percentage of per-protocol subjects who develop titers of ≥ 1:40 as determined by PRNT80 after WEE vaccination at each scheduled time point for which blood samples are drawn and over the entire study period to study completion.

SECONDARY OUTCOMES:
Geometric mean of PRNT80 titers | Up to 5 years
  The geometric mean PRNT80 titers of per-protocol subjects at each scheduled time point for which blood samples are drawn and over the entire study period to study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Cardile, DO, Principal Investigator — US Army Medical Research Institute of Infectious Diseases
Locations (1):
- Special Immunizations Program, USAMRIID, Fort Deterick, Maryland, United States